CLINICAL TRIAL: NCT02388802
Title: The First Human Clinical Trial of Uterine Transplantation in the United Kingdom
Brief Title: Human Clinical Trial of Uterine Transplantation in the United Kingdom
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Womb Transplant UK (Other)
Collaborators: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2015-02-12; First posted 2015-03-17 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Infertility
Keywords: Infertility; Transplant; IVF; Hysterectomy; Absolute uterine infertility
MeSH Terms: conditions — Infertility | interventions — Oocyte Retrieval; Freezing; Immunosuppressive Agents; Fertilization in Vitro; Cesarean Section

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Uterine transplant (Experimental): 10 patients will be appropriately selected to undergo oocyte retrieval and freezing. Subsequently deceased donor allograft excision will take place prior to uterine transplantation. Immunosuppressive agents will be used to optimise graft success until successful In-vitro fertilisation and subsequent delivery by Caesarean Section
  Interventions: Procedure: Oocyte retrieval and freezing; Procedure: Deceased Donor Allograft Excision; Procedure: Uterine Transplantation; Drug: Immunosuppressive Agents; Procedure: In-vitro fertilisation; Procedure: Caesarean Section

INTERVENTIONS:
Procedure: Oocyte retrieval and freezing — 10 Patients will undergo oocyte retrieval and freezing
Procedure: Deceased Donor Allograft Excision — Appropriately matched uterine transplant allografts will be excised from deceased donors
  Other Names: Cadaveric Donor Allograft Excision
Procedure: Uterine Transplantation — Following egg freezing the patients will undergo uterine transplant from deceased donors
  Other Names: Womb Transplant
Drug: Immunosuppressive Agents — Patients will be appropriately immunosuppressed, whilst being closely monitored clinically, radiologically and immunologically.
  Other Names: Immunosuppressives
Procedure: In-vitro fertilisation — 12 months after successful transplantation,the patients will undergo IVF
  Other Names: IVF
Procedure: Caesarean Section — Following successful conception and antenatal period, the babies will be born by Caesarean Section

SUMMARY:
Ten patients will undergo uterine transplantation.

DETAILED DESCRIPTION:
Ten patients that will be appropriately selected using a variety of physical and psychological assessments. The selected patients will undergo egg retrieval and subsequent freezing of embryos to enable IVF treatment following transplantation. Following uterine transplantation, using deceased donor allografts, the patients will be closely monitored for 12 months clinically, radiologically and immunologically until embryo transfer. Following successful embryo transfer the patients will continue to be monitored antenatally until they are delivered by Caesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Between 18-36 years of age
* Absolute Uterine factor infertility

Exclusion Criteria:

* Poor ovarian reserve - Unsuccessful oocyte retrieval
* No intercurrent significant medical or psychiatric co-morbidities
* Previous oncology patients <5 years in remission
* Outside of age range
* Normal BMI

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-01; Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Transplant success | 12 months
  Efficacy as measured by successful graft transplantation with no clinical, immunological or radiological signs of graft rejection within the first 12 months post-operatively.

SECONDARY OUTCOMES:
Pregnancy rate | 24 months
  Efficacy as measured by the number of patients successful of conception by IVF
Live birth rate | 36 months
  Efficacy as measured by the number of live births following successful conception

CONTACTS AND LOCATIONS:
Overall Officials: Richard Smith, FRCOG, MD, Principal Investigator — Imperial NHS Healthcare Trust

REFERENCES:
- [Derived] Jones BP, Vali S, Kasaven LS, Mantrali I, Saso S, Bracewell-Milnes T, Nicopoullos J, Thum MY, Diaz-Garcia C, Quiroga I, Yazbek J, Smith JR. INvestigational Study Into Transplantation of the Uterus (INSITU): a cross-sectional survey among women with uterine factor infertility in the UK assessing background, motivations and suitability. BMJ Open. 2023 Dec 9;13(12):e073517. doi: 10.1136/bmjopen-2023-073517. PMID 38070921